CLINICAL TRIAL: NCT01185340
Title: A Randomized Placebo-Controlled, Double-Blind Study of LY2216684 Flexible-Dose 12 to 18 mg Once Daily as Adjunctive Treatment for Patients With Major Depressive Disorder Who Are Partial Responders to Selective Serotonin Reuptake Inhibitor Treatment
Brief Title: A Study in Participants With Major Depressive Disorder Who Are Partial Responders to Selective Serotonin Reuptake Inhibitor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12183; H9P-MC-LNBR (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder
Keywords: Depression; MDD
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2216684 + SSRI (Experimental): LY2216684: flexible dose of 12 or 18 milligrams (mg), administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Prior to entering the Adjunctive Treatment (AT) Phase, participants completed a 3-week Confirmation (CF) Phase where they received placebo (administered orally, QD) adjunctive to their SSRI. After the CF Phase, and after randomization criteria were met, participants were randomized to the LY2216684 treatment arm.
  For the first 2 weeks of the AT Phase, participants received a starting dose of 12 mg QD. Then, based on efficacy and tolerability, the dose could be increased to 18 mg QD over the next 6 weeks. Participants who had their dose increased to 18 mg QD could have had their dose decreased to 12 mg QD. Participants who completed the AT Phase or discontinued early had the option to enter the Discontinuation (DC) Phase.
  During the 1-week abrupt DC Phase, participants maintained their SSRI treatment.
  Interventions: Drug: LY2216684; Drug: Placebo; Drug: SSRI
- Placebo + SSRI (Placebo Comparator): Placebo: Administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Prior to entering the Adjunctive Treatment (AT) Phase, participants completed a 3-week Confirmation (CF) Phase where they received placebo (administered orally, QD) adjunctive to their SSRI. After the CF Phase, and after randomization criteria were met, participants were randomized to the placebo treatment arm.
  During the AT Phase, participants received placebo (administered orally, QD) adjunctive to their SSRI for 8 weeks. Participants who completed the AT Phase or discontinued early had the option to enter the Discontinuation (DC) Phase.
  During the 1-week abrupt DC Phase, participants maintained their SSRI treatment.
  Interventions: Drug: Placebo; Drug: SSRI

INTERVENTIONS:
Drug: LY2216684
  Other Names: Edivoxetine
  Arms: LY2216684 + SSRI
Drug: Placebo
Drug: SSRI — Participants should have been on their SSRI for at least 6 weeks prior and were to continue on their stable dose throughout the study
  Other Names: selective serotonin reuptake inhibitor

SUMMARY:
The primary objective of this study is to assess whether LY2216684 12 milligrams (mg) or 18 mg flexible dose once daily is superior to placebo once daily in the adjunctive treatment of participants with major depressive disorder (MDD) who are partial responders to their selective serotonin reuptake inhibitor (SSRI) treatment.

DETAILED DESCRIPTION:
Following the Confirmation (CF) Phase, participants were randomized to adjunctive LY2216684 or adjunctive placebo if they had <25% improvement in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score over the past 3 weeks and a current MADRS total score ≥14. Participants who did not meet criteria received adjunctive placebo to preserve the blind.

ELIGIBILITY:
Inclusion Criteria:

* Women of child-bearing potential may participate but must test negative for pregnancy at the time of study entry; both women/men agree to use a reliable method of birth control
* Are being treated with one of the following selective serotonin reuptake inhibitors (SSRIs): escitalopram, citalopram, sertraline, fluoxetine, paroxetine, or fluvoxamine; for at least 6 weeks prior to investigational product dispensing with at least the last 4 weeks at a stable, optimized dose
* Drug and dosage should be within the labeling guidelines for the specific country
* Meet criteria for major depressive disorder (MDD), as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision® (DSM-IV-TR) criteria
* Meet criteria for partial response, as defined by investigator's opinion that the participant has experienced a minimal clinically meaningful improvement with SSRI
* Have a GRID 17-Item Hamilton Depression Rating Scale (GRID-HAMD17) total score greater than or equal to 16 at screening
* Have less than or equal to 75% improvement on the current SSRI at screening determined by the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH-ATRQ)

Exclusion Criteria:

* Have had or currently have any additional ongoing DSM-IV-TR Axis 1 condition other than major depression within 1 year of screening
* Have had any anxiety disorder that was considered a primary diagnosis within the past year (including panic disorder, obsessive-compulsive disorder [OCD], post-traumatic stress disorder [PTSD], generalized anxiety disorder [GAD], and social phobia, but excluding specific phobias)
* Have a current or previous diagnosis of a bipolar disorder, schizophrenia, or other psychotic disorder
* Have a history of substance abuse and/or dependence within the past year (drug categories defined by DSM-IV-TR), not including caffeine and nicotine
* Have an Axis II disorder that, in the judgment of the investigator, would interfere with compliance with protocol
* Unstable medical conditions that contraindicate the use of LY2216684
* Have any diagnosed medical condition that could be exacerbated by noradrenergic agents, including unstable hypertension, unstable heart disease, tachycardia, tachyarrhythmia, narrow-angled glaucoma, history of urinary hesitancy or retention
* Use of excluded concomitant or psychotropic medication other than SSRI
* Have initiated or discontinued hormone therapy within the 3 months prior to enrollment
* History of treatment-resistant depression as shown by lack of response of the current depressive episode to 2 or more adequate courses of antidepressant therapy at a clinically appropriate dose for at least 4 weeks or, in the judgment of the investigator, the participant has treatment-resistant depression
* Have a lifetime history of vagal nerve stimulation (VNS), transcranial magnetic stimulation (TMS), or psychosurgery
* Have received electroconvulsive therapy (ECT) in the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1056 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (49):
- United States (20):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden Grove, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oakland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Temecula, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boca Raton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Bay Village, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oakland Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marlton, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Media, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herndon, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
- Australia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Everton Park, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Hill, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankston, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malvern, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Victoria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Diest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mont-Godinne
- Germany (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Saarow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bochum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cham
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hattingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nuremberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prien am Chiemsee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Schwerin
- Sweden (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gothenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Solna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
- United Kingdom (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bexhill-on-Sea, East Sussex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glasgow, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesterfield

REFERENCES:
- [Derived] Stauffer VL, Liu P, Goldberger C, Marangell LB, Nelson C, Gorwood P, Fava M. Is the Noradrenergic Symptom Cluster a Valid Construct in Adjunctive Treatment of Major Depressive Disorder? J Clin Psychiatry. 2017 Mar;78(3):317-323. doi: 10.4088/JCP.15m09972. PMID 27685842
- [Derived] Ball SG, Ferguson MB, Martinez JM, Pangallo BA, Nery ES, Dellva MA, Sparks J, Zhang Q, Liu P, Bangs M, Goldberger C. Efficacy outcomes from 3 clinical trials of edivoxetine as adjunctive treatment for patients with major depressive disorder who are partial responders to selective serotonin reuptake inhibitor treatment. J Clin Psychiatry. 2016 May;77(5):635-42. doi: 10.4088/JCP.14m09619. PMID 27035159

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The first 3 weeks of the study was a double-blind Confirmation Phase during which participants continued to receive their SSRI with adjunctive placebo. If randomization criteria were met, participants were randomized to adjunctive LY2216684 or adjunctive placebo. If criteria were not met, participants continued on placebo to maintain the blind.
Groups:
- Placebo + SSRI (Pre-randomized Participants): Placebo: Administered orally, once daily for 3 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
- LY2216684 + SSRI (Randomized Participants): LY2216684: 12 or 18 milligrams (mg), administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
- Placebo + SSRI (Randomized Participants); Placebo + SSRI (Non-randomized Participants): Placebo: Administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
Period: Confirmation (CF) Phase, 3 Weeks
Arm/Group | Placebo + SSRI (Pre-randomized Participants) | LY2216684 + SSRI (Randomized Participants) | Placebo + SSRI (Randomized Participants) | Placebo + SSRI (Non-randomized Participants)
Started | 1056 | 0 | 0 | 0
Entered Discontinuation (DC) Phase | 18 (Participants who discontinued the CF Phase early had the option to enter the DC Phase.) | 0 | 0 | 0
Completed | 968 (Participants who completed the CF Phase entered the Adjunctive Treatment (AT) Phase.) | 0 | 0 | 0
Not Completed | 88 | 0 | 0 | 0
Not completed — Adverse Event | 24 | 0 | 0 | 0
Not completed — Lack of Efficacy | 6 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 16 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 32 | 0 | 0 | 0
Not completed — Sponsor Decision | 3 | 0 | 0 | 0
Period: Adjunctive Treatment (AT) Phase, 8 Weeks
Arm/Group | Placebo + SSRI (Pre-randomized Participants) | LY2216684 + SSRI (Randomized Participants) | Placebo + SSRI (Randomized Participants) | Placebo + SSRI (Non-randomized Participants)
Started | 0 | 230 | 219 | 519
Entered Discontinuation (DC) Phase | 0 | 206 (Participants who completed the AT Phase or discontinued early had the option to enter the DC Phase.) | 204 (Participants who completed the AT Phase or discontinued early had the option to enter the DC Phase.) | 483 (Participants who completed the AT Phase or discontinued early had the option to enter the DC Phase.)
Completed | 0 | 195 | 186 | 458
Not Completed | 0 | 35 | 33 | 61
Not completed — Adverse Event | 0 | 13 | 8 | 13
Not completed — Lack of Efficacy | 0 | 4 | 7 | 4
Not completed — Lost to Follow-up | 0 | 4 | 5 | 7
Not completed — Physician Decision | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 5 | 2 | 5
Not completed — Withdrawal by Subject | 0 | 8 | 8 | 24
Not completed — Sponsor Decision | 0 | 0 | 3 | 7

BASELINE CHARACTERISTICS:
Population: Participants who completed the Confirmation (CF) Phase and were randomized to adjunctive LY2216684 or adjunctive placebo or who did not met randomization criteria and continued on placebo to maintain the blind.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2216684 + SSRI (Randomized Participants) | Placebo + SSRI (Randomized Participants) | Placebo + SSRI (Non-randomized Participants) | Total
Number analyzed (Participants) | 230 | 219 | 519 | 968
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.29 (11.90) | 48.44 (11.39) | 47.39 (12.68) | 47.84 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 145 | 354 | 654
  Male | 75 | 74 | 165 | 314
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 12 | 31 | 62
  Not Hispanic or Latino | 164 | 158 | 370 | 692
  Unknown or Not Reported | 47 | 49 | 118 | 214
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 3 | 3
  Asian | 2 | 1 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 31 | 53 | 101
  White | 207 | 185 | 457 | 849
  More than one race | 4 | 2 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 93 | 89 | 195 | 377
  Belgium | 7 | 4 | 13 | 24
  Austria | 10 | 10 | 25 | 45
  Australia | 22 | 20 | 84 | 126
  Germany | 58 | 63 | 95 | 216
  United Kingdom | 19 | 15 | 30 | 64
  Sweden | 21 | 18 | 77 | 116

OUTCOME MEASURES:

1. Primary Outcome: Change From Randomization to Week 8 in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: All randomized participants who have non-missing values at the time of randomization and at least one post-randomization value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- LY2216684 + SSRI: LY2216684: 12 or 18 milligrams (mg), administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
- Placebo + SSRI: Placebo: Administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 225 | 217
units on a scale | -8.73 (0.55) | -8.49 (0.57)
Statistical Analysis 1: Comparison: LY2216684 + SSRI vs Placebo + SSRI; Test type: Superiority or Other; p = 0.751, Mixed Models Analysis

2. Secondary Outcome: Change From Randomization to Week 8 in Sheehan Disability Scale (SDS) Global Functional Impairment Score
Description: The Sheehan Disability Scale (SDS) was completed by the participant and used to assess the effect of the participant's symptoms on their work (Item 1), social (Item 2), and family life (Item 3). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. The Global Functional Impairment Score is the sum of the 3 items, and scores ranged from 0 to 30 with higher values indicating greater disruption in the participant's work life (work/school impairment score), social life (social life/leisure activities impairment score), and family life (family life/home responsibilities impairment score). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 218 | 208
units on a scale | -4.50 (0.47) | -4.38 (0.48)

3. Secondary Outcome: Change From Randomization to Week 8 in Fatigue Associated With Depression (FAsD) Impact Subscale Score
Description: The Fatigue Associated with Depression (FAsD) is a participant-rated scale with a total of 13 items. Six of the 13 items ask how often participants experience different aspects of fatigue with responses from 1 (never) to 5 (always). Seven of the 13 items ask how often fatigue impacts various aspects of the participant's lives with responses from 1 (not at all) to 5 (very much). The impact subscale score was derived by taking the mean of Items 7 through 13 (applicable items only). Item 12 applied only to participants with a spouse or significant other, and Item 13 applied to participants who had a job or who went to school. The FAsD impact subscale score ranges from 1 to 5. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline subscale score, treatment-by-visit, and baseline subscale score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 218 | 209
units on a scale | -0.69 (0.06) | -0.59 (0.07)

4. Secondary Outcome: Probability of Participants Achieving a Montgomery-Asberg Depression Rating Scale (MADRS) Total Score of Less Than or Equal to 10 at Week 8
Description: A Montgomery-Asberg Depression Rating Scale (MADRS) total score of less than or equal to 10 was defined as remission criteria. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). A categorical repeated measures analysis modeled the probability of remission at each visit, and the estimated probabilities were adjusted for treatment, visit, baseline MADRS total score, and treatment-by-visit.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: probability
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 225 | 217
probability | 0.313 (0.034) | 0.251 (0.032)

5. Secondary Outcome: Percentage of Participants Achieving a Montgomery-Asberg Depression Rating Scale (MADRS) Total Score of Less Than or Equal to 10 for at Least 2 Consecutive Measurements, Including the Participant's Last Measurement
Description: A Montgomery-Asberg Depression Rating Scale (MADRS) total score of less than or equal to 10 for at least 2 consecutive measurements, including the participant's last measurement was defined as remission criteria at last 2 consecutive visits. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Percentage of participants was calculated by dividing the number of participants who meet criteria for remission at last 2 consecutive visits by the total number of participants analyzed, multiplied by 100%.
Time Frame: Randomization up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 225 | 218
percentage of participants | 20.89 | 17.89

6. Secondary Outcome: Change From Randomization to Week 8 in Hospital and Anxiety and Depression Scale (HADS) Anxiety Subscale Score
Description: The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire with 2 subscales: anxiety and depression. Each item was rated on a 4-point scale (0-3), giving maximum scores of 21 for anxiety and depression subscale. Scores of 11 or more on either subscale were considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7 represent 'normal'. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline subscale score, treatment-by-visit, and baseline subscale score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 224 | 217
units on a scale | -2.20 (0.22) | -1.78 (0.23)

7. Secondary Outcome: Probability of Participants Who Have a Greater Than or Equal to 50 Percent Improvement in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Week 8
Description: A greater than or equal to 50 percent improvement (that is, a decrease from baseline) in the Montgomery-Asberg Depression Rating Scale (MADRS) total score was defined as response criteria. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). A categorical repeated measures analysis modeled the probability of response at each visit, and the estimated probabilities were adjusted for treatment, visit, baseline MADRS total score, and treatment-by-visit.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: probability
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 225 | 217
probability | 0.357 (0.034) | 0.352 (0.034)

8. Secondary Outcome: Change From Randomization to Week 8 in The Hospital Anxiety and Depression Scale (HADS) Depression Subscale Score
Description: as for outcome 6
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 224 | 217
units on a scale | -2.82 (0.27) | -2.64 (0.27)

9. Secondary Outcome: Change From Randomization to Week 8 in Montgomery-Asberg Depression Rating Scale (MADRS) Individual Items
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline item score, treatment-by-visit and baseline item score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 225 | 217
units on a scale
  Apparent Sadness | -1.10 (0.09) | -1.26 (0.09)
  Reported Sadness | -1.17 (0.09) | -1.19 (0.09)
  Inner Tension | -0.72 (0.08) | -0.71 (0.09)
  Reduced Sleep | -0.83 (0.09) | -0.76 (0.10)
  Reduced Appetite | -0.54 (0.08) | -0.72 (0.08)
  Concentration Difficulties | -1.07 (0.09) | -0.82 (0.09)
  Lassitude | -1.11 (0.09) | -0.98 (0.09)
  Inability to Feel | -1.17 (0.09) | -1.08 (0.09)
  Pessimistic Thoughts | -0.88 (0.08) | -0.77 (0.08)
  Suicidal Thoughts | -0.23 (0.05) | -0.24 (0.05)

10. Secondary Outcome: Change From Randomization to Week 8 in Clinical Global Impressions of Severity (CGI-S)
Description: Clinical Global Impression - Severity (CGI-S) measures severity of depression at the time of assessment compared with the start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 224 | 217
units on a scale | -1.08 (0.08) | -1.02 (0.08)

11. Secondary Outcome: Change From Randomization to Week 8 in Fatigue Associated With Depression (FAsD) Average Score and Experience Subscale Score
Description: The Fatigue Associated with Depression (FAsD) is a participant-rated scale with a total of 13 items. Six of the 13 items ask how often participants experience different aspects of fatigue with responses from 1 (never) to 5 (always). Seven of the 13 items ask how often fatigue impacts various aspects of the participant's lives with responses from 1 (not at all) to 5 (very much). The experience subscale score was derived by taking the mean of Items 1 through 6, and the average score was the mean of Items 1 through 13 (derived by taking the mean of all applicable items for each participant). Item 12 applied only to participants with a spouse or significant other, and Item 13 applied to participants who had a job or who went to school. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 217 | 210
units on a scale
  FAsD average score: number analyzed (Participants) | 217 | 209
  FAsD average score | -0.62 (0.06) | -0.55 (0.06)
  FAsD experience subscale score | -0.57 (0.06) | -0.50 (0.06)

12. Secondary Outcome: Change From Randomization to Week 8 in Sheehan Disability Scale (SDS) Items
Description: The Sheehan Disability Scale (SDS) was completed by the participant and used to assess the effect of the participant's symptoms on their work (work/school impairment score), social life (social life/leisure activities impairment score), and family life (family life/home responsibilities impairment score). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline item score, treatment-by-visit, and baseline item score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 218 | 209
units on a scale
  Work impairment score: number analyzed (Participants) | 138 | 135
  Work impairment score | -1.41 (0.22) | -1.20 (0.22)
  Social life impairment score | -1.64 (0.17) | -1.53 (0.17)
  Family life impairment score: number analyzed (Participants) | 218 | 208
  Family life impairment score | -1.56 (0.17) | -1.53 (0.17)

13. Secondary Outcome: Change From Randomization to Week 8 in the Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF)
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) is a self-administered, 16-item questionnaire measuring degree of enjoyment and satisfaction experienced in various areas of daily life during the past week on a 5-point Likert scale (1=very poor and 5=very good). The total raw score is the sum of Items 1 to 14 and ranges from 14 to 70. The raw scores are converted to and expressed as the percentage of the maximum possible score. Higher scores indicate higher levels of enjoyment/satisfaction. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of the maximum possible score
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 218 | 208
percentage of the maximum possible score | 10.37 (1.09) | 9.30 (1.12)

14. Secondary Outcome: Change From Randomization to Week 8 in the EuroQol Questionnaire-5 Dimension (EQ-5D)
Description: The EQ-5D Visual Analog Scale is a generic, multidimensional, health-related, quality-of-life instrument. Overall health state score is self-reported using a visual analogue scale, marked on a scale of 0 to 100 with 0 representing worst imaginable health state and 100 representing best imaginable health state. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 216 | 209
units on a scale | 10.367 (1.218) | 9.644 (1.252)

15. Secondary Outcome: Percentage of Participants With Treatment-emergent Suicidal Ideation and Behaviors Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) captured occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation was defined as a "yes" answer to any 1 of 5 suicidal ideation questions, which included a wish to be dead and 4 different categories of active suicidal ideation. Suicidal behavior was defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation and behavior are defined as treatment-emergent (TE) if not present at baseline. Percentage of participants was calculated by dividing the number of participants with suicide-related TE events by the total number of participants at risk, multiplied by 100%. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Event module.
Time Frame: Randomization up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 224 | 218
percentage of participants
  TE suicidal ideation | 4.46 | 5.96
  TE suicidal behavior: number analyzed (Participants) | 206 | 193
  TE suicidal behavior | 0.00 | 0.52

16. Secondary Outcome: Change From Randomization to Week 8 in Arizona Sexual Experiences (ASEX) Scale
Description: The Arizona Sexual Experiences (ASEX) scale was used to assess sexual functioning in both males and females. The ASEX total score for the male and female version was calculated as the sum of the responses (rated from 1 [extremely] to 6 [no/never]) of the 5 items of the ASEX scale. Total scores ranged from 5 to 30, with higher scores indicating greater sexual dysfunction. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 214 | 204
units on a scale | -0.92 (0.25) | -0.68 (0.26)

17. Secondary Outcome: Change From Randomization to Week 8 in Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ)
Description: The Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) is a 7-item participant-rated questionnaire pertaining to a participant's cognitive and physical well-being. It assesses motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each item was scored on a 6-point scale ranging from 1 (greater than normal) to 6 (totally absent). Total scores ranged from 7 to 42. Higher scores indicate greater disease severity. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 218 | 210
units on a scale | -4.12 (0.39) | -3.68 (0.40)

18. Secondary Outcome: Change From Randomization to Week 8 in Blood Pressure
Description: Blood pressure measurements were collected when the participant was in a sitting position. Three measurements of sitting blood pressure collected at approximately 1-minute intervals at every visit were averaged and used as the value for the visit. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline value, treatment-by-visit, and baseline value-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 225 | 217
millimeters of mercury (mmHg)
  Systolic blood pressure | 3.09 (0.67) | 0.27 (0.69)
  Diastolic blood pressure | 4.54 (0.53) | 0.53 (0.54)

19. Secondary Outcome: Change From Randomization to Week 8 in Pulse Rate
Description: Pulse measurements were collected when the participant was in a sitting position. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline value, treatment-by-visit, and baseline value-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 225 | 216
beats per minute (bpm) | 9.64 (0.67) | -1.49 (0.69)

ADVERSE EVENTS:
Time Frame: Confirmation (CF) Phase: Week 0 through Week 3 Adjunctive Treatment (AT) Phase: Week 4 through Week 11 Discontinuation (DC) Phase: The week following completion of the AT Phase (Week 12) or early discontinuation of the CF Phase or AT Phase
Groups:
- Placebo + SSRI (Pre-randomized) - CF Phase: Placebo: Administered orally, once daily for 3 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Includes all enrolled participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-baseline visit during the Confirmation (CF) Phase.
- LY2216684 + SSRI (Randomized) - AT Phase: LY2216684: 12 or 18 milligrams (mg), administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Includes randomized participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-randomization visit during the Adjunctive Treatment (AT) Phase.
- Placebo + SSRI (Randomized) - AT Phase: Placebo: Administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Includes randomized participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-randomization visit during the Adjunctive Treatment (AT) Phase.
- Placebo + SSRI (Non-randomized) - AT Phase: Placebo: Administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Includes all non-randomized participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-randomization visit during the Adjunctive Treatment (AT) Phase.
- Placebo + SSRI (Pre-randomized) - DC Phase: No study drug was administered. Participants were to maintain their selective serotonin reuptake inhibitor (SSRI) treatment at a stable dose for 1 week.
  Includes all enrolled participants who abruptly discontinued placebo after early withdrawal during the Confirmation (CF) Phase and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
- LY2216684 + SSRI (Randomized) - DC Phase: No study drug was administered. Participants were to maintain their selective serotonin reuptake inhibitor (SSRI) treatment at a stable dose for 1 week.
  Includes all randomized participants who abruptly discontinued LY2216684 either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
- Placebo + SSRI (Randomized) - DC Phase: No study drug was administered. Participants were to maintain their selective serotonin reuptake inhibitor (SSRI) treatment at a stable dose for 1 week.
  Includes all randomized participants who abruptly discontinued placebo either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
- Placebo + SSRI (Non-randomized) - DC Phase: No study drug was administered. Participants were to maintain their selective serotonin reuptake inhibitor (SSRI) treatment at a stable dose for 1 week.
  Includes all non-randomized participants who abruptly discontinued placebo either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
Arm/Group | Placebo + SSRI (Pre-randomized) - CF Phase | LY2216684 + SSRI (Randomized) - AT Phase | Placebo + SSRI (Randomized) - AT Phase | Placebo + SSRI (Non-randomized) - AT Phase | Placebo + SSRI (Pre-randomized) - DC Phase | LY2216684 + SSRI (Randomized) - DC Phase | Placebo + SSRI (Randomized) - DC Phase | Placebo + SSRI (Non-randomized) - DC Phase
Serious Adverse Events (participants affected / at risk) | 9/1052 | 7/228 | 7/218 | 12/519 | 1/18 | 2/206 | 4/202 | 4/482
Other Adverse Events (participants affected / at risk) | 270/1052 | 87/228 | 44/218 | 128/519 | 5/18 | 39/206 | 22/202 | 70/482
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + SSRI (Pre-randomized) - CF Phase (N=1052) | LY2216684 + SSRI (Randomized) - AT Phase (N=228) | Placebo + SSRI (Randomized) - AT Phase (N=218) | Placebo + SSRI (Non-randomized) - AT Phase (N=519) | Placebo + SSRI (Pre-randomized) - DC Phase (N=18) | LY2216684 + SSRI (Randomized) - DC Phase (N=206) | Placebo + SSRI (Randomized) - DC Phase (N=202) | Placebo + SSRI (Non-randomized) - DC Phase (N=482)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + SSRI (Pre-randomized) - CF Phase (N=1052) | LY2216684 + SSRI (Randomized) - AT Phase (N=228) | Placebo + SSRI (Randomized) - AT Phase (N=218) | Placebo + SSRI (Non-randomized) - AT Phase (N=519) | Placebo + SSRI (Pre-randomized) - DC Phase (N=18) | LY2216684 + SSRI (Randomized) - DC Phase (N=206) | Placebo + SSRI (Randomized) - DC Phase (N=202) | Placebo + SSRI (Non-randomized) - DC Phase (N=482)
Abdominal discomfort (Gastrointestinal disorders) | 6 (7) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 33 (35) | 9 (9) | 4 (4) | 7 (7) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 54 (56) | 19 (24) | 7 (9) | 16 (17) | 2 (2) | 4 (4) | 5 (5) | 10 (10)
Vomiting (Gastrointestinal disorders) | 7 (7) | 14 (16) | 4 (5) | 7 (7) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 36 (37) | 12 (13) | 11 (12) | 31 (31) | 1 (1) | 2 (2) | 0 (0) | 6 (6)
Dizziness (Nervous system disorders) | 28 (30) | 14 (14) | 6 (6) | 7 (7) | 1 (1) | 3 (3) | 4 (4) | 9 (9)
Headache (Nervous system disorders) | 117 (137) | 26 (35) | 14 (17) | 53 (64) | 3 (3) | 27 (30) | 14 (14) | 47 (53)
Somnolence (Nervous system disorders) | 11 (12) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Tension headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 4 (4) | 4 (5) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 29 (29) | 27 (27) | 2 (2) | 14 (14) | 0 (0) | 4 (4) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days